CLINICAL TRIAL: NCT00081640
Title: Phase I Safety and Acceptability Study of the Investigational Vaginal Microbicide PRO 2000/5 Gel (P)
Brief Title: Safety and Acceptability of PRO 2000 Vaginal Gel in HIV Uninfected Women in India
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 047
Record Dates: First submitted 2004-04-16; First posted 2004-04-19 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2006-11

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Vaginal Microbicide
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: PRO 2000/5 Gel (P)

SUMMARY:
PRO 2000 Gel is designed to be inserted into the vagina to protect women from getting HIV during sex. So far, PRO 2000 Gel has been tested for safety in 136 women from Europe and the United States. This study will evaluate the safety and acceptability of PRO 2000 Gel when used by women in Pune, India. The study will also examine what Indian women and men think about using PRO 2000 Gel.

DETAILED DESCRIPTION:
Topical microbicides are designed to prevent the sexual transmission of HIV and other disease pathogens. PRO 2000/5 Gel (P), or PRO 2000, is a vaginal microbicide that has been evaluated in Phase I safety trials in Europe and the U.S. PRO 2000 Gel is easily manufactured, highly stable, and highly water-soluble. The aqueous gel formulation contains a synthetic carbomer, a lactic acid/lactate buffer, and preservatives. In vitro, PRO 2000 Gel has been shown to suppress infection by herpes viruses, Chlamydia trachomatis, Neisseria gonorrhoeae, and a wide range of HIV-1 isolates. This study will evaluate the safety and acceptability of PRO 2000 Gel in HIV uninfected women in Pune, India. The study is a precursor to a larger Phase II/III study of PRO 2000 Gel.

Participants in this study will be sexually active HIV uninfected women at either low or high risk for HIV infection. Male partners of these women will also be enrolled in the study. Participants will be asked to apply PRO 2000 Gel twice a day for 14 consecutive days between menses and to have vaginal intercourse with a single male partner, using study-provided male condoms, at least twice per week during the two weeks of PRO 2000 Gel use. Participants will have a screening visit, an enrollment visit, and 3 study visits during the two weeks of PRO 2000 Gel use; each visit will last about 1 hour. Study visits will include a medical history, gynecologic exam, blood and urine tests, and product acceptability questionnaires. Colposcopy will be performed three times during the study. Participants will also be asked to complete a Daily Study Record about product use and sexual activity and questionnaires about their willingness to use the product and their perceptions of the product.

Four weeks after using PRO 2000 Gel, participants will be asked to participate in a focus group to discuss product acceptability. Participants' male partners will also be asked to participate in focus groups about product use.

ELIGIBILITY:
Inclusion Criteria for All Female Participants:

* Age 18 to 45
* HIV uninfected
* Regular menstrual cycle of at least 21 days or no menstrual cycle because of long-acting progestin use
* No change in hormonal contraceptive use in the 3 months prior to study entry
* Agree to use acceptable methods of contraception during the study
* Normal Pap smear at screening or in the 3 months prior to study entry
* Sexually active with a single male sexual partner who is eligible for the study
* Agree to abstain from sexual intercourse for 48 hours before the enrollment visit
* Willing to complete Daily Study Records
* Agree to follow study directions about PRO 2000 Gel use and sexual activity during the study

Additional Inclusion Criteria for Female Participants at Higher Risk for HIV Infection:

* Sexually transmitted disease (STD) in the 3 months prior to study entry
* Current male partner has had an STD in the 3 months prior to study entry

Inclusion Criteria for Male Partners of Female Participants:

* Age 18 years or older
* HIV uninfected
* No STD symptoms at study entry
* Agree to abstain from sexual intercourse for 48 hours before the enrollment visit
* Agree to have vaginal intercourse only with partner who is taking part in the study
* Agree to have vaginal intercourse at least twice a week while in the study and to use study provided male condoms

Exclusion Criteria for All Female Participants:

* Menopausal
* Breastfeeding
* Used non-therapeutic intravenous drugs within 1 year of study
* Currently pregnant or have been pregnant in the 3 months prior to study entry
* Serious liver, kidney, or blood abnormalities
* Urinary tract infection as determined by positive urine culture
* Genital abnormality
* History of adverse reaction to anticoagulants
* History of sensitivity or allergy to latex
* Used any spermicide or spermicidally lubricated condom in the week prior to study entry
* Participated in any investigational drug trial in 30 days prior to study entry
* Used an intrauterine contraceptive device in the 3 months prior to study entry
* Abnormal Pap smear in the 3 months prior to study entry
* Gynecological surgery in the 3 months prior to study entry
* Breakthrough menstrual bleeding in the 3 months prior to study entry
* Vaginal bleeding during or following intercourse in the 3 months prior to study entry

Additional Exclusion Criteria for Female Participants at Low Risk for HIV Infection:

* STD or pelvic inflammatory disease in the 3 months prior to study entry
* Current male partner has had an STD in the 3 months prior to study entry
* Current male partner has injected non-therapeutic drugs in the 3 months prior to study entry
* Signs on pelvic exam consistent with an STD other than bacterial vaginosis

Exclusion Criteria for Male Partners of Female Participants

* History of adverse reaction to latex
* Refuse examination or treatment for an STD or STD symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120

CONTACTS AND LOCATIONS:
Overall Officials: Smita N. Joshi, MBBS, Study Chair — National AIDS Research Institute (Pune, India); Steven J. Reynolds, MD, FRCP(C), Study Chair — Johns Hopkins University Department of Medicine

REFERENCES:
- [Background] Morrow K, Rosen R, Richter L, Emans A, Forbes A, Day J, Morar N, Maslankowski L, Profy AT, Kelly C, Abdool Karim SS, Mayer KH. The acceptability of an investigational vaginal microbicide, PRO 2000 Gel, among women in a phase I clinical trial. J Womens Health (Larchmt). 2003 Sep;12(7):655-66. doi: 10.1089/154099903322404302. PMID 14583106
- [Background] Tabet SR, Callahan MM, Mauck CK, Gai F, Coletti AS, Profy AT, Moench TR, Soto-Torres LE, Poindexter III AN, Frezieres RG, Walsh TL, Kelly CW, Richardson BA, Van Damme L, Celum CL. Safety and acceptability of penile application of 2 candidate topical microbicides: BufferGel and PRO 2000 Gel: 3 randomized trials in healthy low-risk men and HIV-positive men. J Acquir Immune Defic Syndr. 2003 Aug 1;33(4):476-83. doi: 10.1097/00126334-200308010-00008. PMID 12869836
- [Background] Mayer KH, Karim SA, Kelly C, Maslankowski L, Rees H, Profy AT, Day J, Welch J, Rosenberg Z; HIV Prevention Trials Network (HPTN) 020 Protocol Team. Safety and tolerability of vaginal PRO 2000 gel in sexually active HIV-uninfected and abstinent HIV-infected women. AIDS. 2003 Feb 14;17(3):321-9. doi: 10.1097/00002030-200302140-00005. PMID 12556685
- [Background] Trager RS. Microbicides. Raising new barriers against HIV infection. Science. 2003 Jan 3;299(5603):39. doi: 10.1126/science.299.5603.39. No abstract available. PMID 12511630
- [Result] Smita J, Soma D, Beverly B, Albert P, JoAnn K, Fang G, Missy C, Lydia ST, Anjali P, Arun R, Sanjay M, Steven J R; HIV Prevention Trial Network (HPTN) 047 Protocol Team. Phase I safety study of 0.5% PRO 2000 vaginal Gel among HIV un-infected women in Pune, India. AIDS Res Ther. 2006 Feb 20;3:4. doi: 10.1186/1742-6405-3-4. PMID 16504023